CLINICAL TRIAL: NCT06967324
Title: GRACE - Graduated Response for Advanced COPD With Enhanced Support
Acronym: GRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Kirstine Skov Benthien, Senior Researcher, associate professor, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-25009646
Record Dates: First submitted 2025-05-12; First posted 2025-05-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; palliative care; cross-sectoral
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cross-sectoral stepped care with systematic needs assessment, advance care planning and virtual conferences
  Interventions: Other: Stepped care; Other: Usual Care
- Control (Active Comparator): Care as usual at the outpatient respiratory clinic
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Stepped care — Graduated palliative cross-sectoral care
  Arms: Intervention
Other: Usual Care — Usual care at the outpatient respiratory clinic

SUMMARY:
The aim of this study is to explore the feasibility and potential for a positive impact of a graduated response for advanced COPD with Enhanced Support. The study is a randomized controlled trial of:

* systematic needs assessment
* advance care planning
* crossectoral virtual conferences. Researchers will compare quality of life and healthcare use of the intervention group with a control group that will be assessed for intervention need at the last follow-up.

DETAILED DESCRIPTION:
The current study is a non-blinded randomized controlled pilot trial. The control group will be offered treatment as usual whereas the intervention group will be allocated to the GRACE model of care. In total, 100 patients and their caregivers will be included. The patients are all community dwelling and attached to the Outpatient Respiratory Medicine Clinic at Hvidovre Hospital. The patients will be randomized by block randomization to intervention and control group with a ratio of 1:1. Furthermore, the patients will be stratified according to which municipality they belong to, to ensure we gather feasibility data from two municipalities. The control group will be offered to be assessed for their eligibility for palliative care through the existing visitation conference at the end of the trial period. Endpoints include: Patient-reported (quality of life, anxiety and depression, self-efficacy), caregiver-reported ( caregiver burden, anxiety and depression, well-being) and patient healthcare use.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Exacerbation within the last year
* Living in Høje Taastrup or Copenhagen
* Cognitively relevant
* ICECAP-SCM at least two scores of:

  1. 1, 2
  2. 1, 2
  3. 1, 2
  4. 1, 2
  5. 1, 2, 3
  6. 1, 2
  7. 1, 2

Exclusion Criteria:

* Dementia
* Psychosis
* Substance abuse
* Hearing or speech impairment
* Cancer
* Receiving specialized palliative care or other similar interventions
* Immediately dying

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
ICECAP-SCM | 6 months

SECONDARY OUTCOMES:
ICECAP-SCM | 3 months
ICECAP-SCM | 9 months
ICECAP-SCM | 12 months
HADS | 3
  Anxiety and depression
HADS | 6
  Anxiety and depression
HADS | 9 months
  Anxiety and depression
HADS | 12 months
  Anxiety and depression
GSE | 3 months
  General self-efficacy scale
GSE | 6 months
  General self-efficacy scale
GSE | 9 months
  General self-efficacy scale
GSE | 12 months
  General self-efficacy scale
Hospital admissions | 3 months
  * Proportion of patients with any hospital admission
  * Mean number of admissions per patient
  * Bed days
Hospital admissions | 6 months
  * Proportion of patients with any hospital admission
  * Mean number of admissions per patient
  * Bed days
Hospital admissions | 9 months
  * Proportion of patients with any hospital admission
  * Mean number of admissions per patient
  * Bed days
Hospital admissions | 12 months
  * Proportion of patients with any hospital admission
  * Mean number of admissions per patient
  * Bed days
Healthcare use, municipality | 3 months
Healthcare use, municipality | 6 months
Healthcare use, municipality | 9 months
Healthcare use, municipality | 12 months
Healthcare use, hospital | 3 months
Healthcare use, hospital | 6 months
Healthcare use, hospital | 9 months
Healthcare use, hospital | 12 months
Healthcare use, general practice | 3 months
Healthcare use, general practice | 6 months
Healthcare use, general practice | 9 months
Healthcare use, general practice | 12 months
Survival | 12 months
SF12 | 3 months
  Health-related quality of life
SF12 | 6 months
  Health-related quality of life
SF12 | 9 months
  Health-related quality of life
SF12 | 12 months
  Health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine Benthien, Ph.d., Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital - Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided